CLINICAL TRIAL: NCT03915873
Title: Assessing the Bleeding Severity in Type I Von Willebrand Patients Using the International Society on Thrombosis and Hemostasis Bleeding Assessment Tool ( ISTH-BAT) Questionnaire
Brief Title: Evaluation of Bleeding Score in Egyptian Patients With vWD Type I and Correlate it With Laboratory Parameters
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shery nabil Hennes abdl-sayed, principal investigator, Assiut University
Other Study IDs: BS in VWD
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Von Willebrand Disease, Type 1
Keywords: von willebrand; egyptian; questionnaire
MeSH Terms: conditions — von Willebrand Disease, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vWB patients
  Interventions: Diagnostic Test: The von Willebrand Antigen level
- control

INTERVENTIONS:
Diagnostic Test: The von Willebrand Antigen level — blood sample
  Groups: vWB patients

SUMMARY:
Applying the ISTH-BAT questionnaire on Egyptian patients with type I VWD aiming to correlate the BS with the laboratory findings

DETAILED DESCRIPTION:
The clinical phenotype of the disease is variable and tends to be mild in type 1 vWD, whereas it shows serious bleeding manifestations in types 2 and 3. Overall, the symptoms reported in vWD include easy bruising, epistaxis, gastrointestinal bleeding, excessive menstrual bleeding, postpartum haemorrhage, and excessive bleeding after surgical operation and minor wounds.However, A distinctive bleeding history is a prerequisite for the diagnosis of any bleeding disorder and should guide further laboratory investigations In an attempt to standardize the diagnostic criteria of VWD, a bleeding questionnaire and a bleeding score were developed The combination of a standardized bleeding questionnaire and a well-defined interpretation grid (for the computation of the final (BS) has been referred to as a Bleeding Assessment Tool (BAT).

ELIGIBILITY:
Inclusion Criteria:

* type 1 vWD patients
* healthy subjects with no known problem with bleeding or bruising were also recruited

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: type 1 von willebrand egyptian patients
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
the International Society on Thrombosis and Hemostasis-Bleeding Assessment Tool (ISTH-BAT) | one year
  Questionnaire minimum score ranges from 0 to 10 whereas maximum score ranges from 20 to 30